CLINICAL TRIAL: NCT01609725
Title: Impact of Periodontal Therapy in Flow-mediated Dilation and Serum Levels of Cardiovascular Risk Biomarkers in Coronary Artery Disease Patients: 12 Months Randomized Controlled Trial
Brief Title: Periodontal Therapy in Coronary Artery Patients
Acronym: PerioCardio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Alex Nogueira Haas, Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HCPA110146
Record Dates: First submitted 2012-05-29; First posted 2012-06-01 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Cardiovascular Diseases; Atheroma; Coronary Artery Disease
Keywords: Coronary artery disease; C reactive protein; Periodontitis; Periodontal therapy; Flow-mediated dilation
MeSH Terms: conditions — Cardiovascular Diseases; Plaque, Atherosclerotic; Coronary Artery Disease; Periodontitis | interventions — Dental Scaling; Root Planing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comprehensive treatment (Experimental): Test treatment group
  Interventions: Device: Subgingival scaling and root planing
- Community treatment (Other): Control treatment group
  Interventions: Device: Oral prophylaxis

INTERVENTIONS:
Device: Subgingival scaling and root planing — Oral hygiene instruction and motivation will be provided altogether with scaling and root planing of all teeth affected by periodontitis under local anesthesia
  Arms: Comprehensive treatment
Device: Oral prophylaxis — One session of supraginigval calculus removal
  Arms: Community treatment

SUMMARY:
Gingival inflammation has been associated with cardiovascular diseases, including heart attack and stroke, because of elevation of blood risk markers such as cholesterol, glucose and C reactive protein. The treatment of gingival diseases decreases the concentration of these risk factors in the blood of cardiovascular patients.

ELIGIBILITY:
Inclusion Criteria:

* 35 years and older
* coronary artery disease
* more than 10 teeth
* chronic periodontitis defined as 2 non-adjacent teeth with probing depth 5+mm and periodontal attachment loss 4+mm

Exclusion Criteria:

* use of antibiotics in the last 6 months
* periodontal therapy in the last 12 months

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2012-01; Primary Completion 2016-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Changes in C reactive protein | Baseline, 3, 6 and 12 months
Changes in flow-mediated dilation | Baseline, 1, 3 and 6 months

SECONDARY OUTCOMES:
Changes in Interleukin 1B concentrations | Baseline, 3, 6, 12 months
Changes in TNF alpha | Baseline, 3, 6, 12 months
Changes in Interleukin 8 | Baseline, 3, 6, 12 months
Changes in Interleukin 6 | Baseline, 3, 6, 12 months
Changes in Cholesterol | Baseline, 3, 6, 12 months
Changes in Glycated hemoglobin | Baseline, 3, 6, 12 months
Changes in LDL/HDL | Baseline, 3, 6, 12 months
Changes in Fibrinogen | Baseline, 3, 6, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alex N Haas, PhD, Study Chair — Federal University of Rio Grande do Sul, Periodontology; Cassiano K Rosing, PhD, Study Chair — Federal University of Rio Grande do Sul, Periodontology; Carisi Polanczyk, PhD, Study Chair — Federal University of Rio Grande do Sul, Cardiology; Eneida RR Rabelo da Silva, PhD, Study Chair — Federal University of Rio Grande do Sul; Marco A Saffi, MS, Principal Investigator — Federal University of Rio Grande do Sul, Cardiology; Cassio Kampits, MS, Principal Investigator — Federal University of Rio Grande do Sul, Periodontology; Ingrid Sanada, MS, Principal Investigator — Federal University of Rio Grande do Sul, Periodontology; Marlon Montenegro, MS, Principal Investigator — Federal University of Rio Grande do Sul, Periodontology; Mariana V Furtado, MS, Study Director — Federal University of Rio Grande do Sul, Cardiology
Locations (1):
- Federal University of Rio Grande do Sul, School of Dentistry and University Hospital, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Ramirez JH, Arce RM, Contreras A. Periodontal treatment effects on endothelial function and cardiovascular disease biomarkers in subjects with chronic periodontitis: protocol for a randomized clinical trial. Trials. 2011 Feb 16;12:46. doi: 10.1186/1745-6215-12-46. PMID 21324167
- [Background] Paraskevas S, Huizinga JD, Loos BG. A systematic review and meta-analyses on C-reactive protein in relation to periodontitis. J Clin Periodontol. 2008 Apr;35(4):277-90. doi: 10.1111/j.1600-051X.2007.01173.x. Epub 2008 Feb 20. PMID 18294231
- [Background] Blaizot A, Vergnes JN, Nuwwareh S, Amar J, Sixou M. Periodontal diseases and cardiovascular events: meta-analysis of observational studies. Int Dent J. 2009 Aug;59(4):197-209. PMID 19774803
- [Background] Lockhart PB, Bolger AF, Papapanou PN, Osinbowale O, Trevisan M, Levison ME, Taubert KA, Newburger JW, Gornik HL, Gewitz MH, Wilson WR, Smith SC Jr, Baddour LM; American Heart Association Rheumatic Fever, Endocarditis, and Kawasaki Disease Committee of the Council on Cardiovascular Disease in the Young, Council on Epidemiology and Prevention, Council on Peripheral Vascular Disease, and Council on Clinical Cardiology. Periodontal disease and atherosclerotic vascular disease: does the evidence support an independent association?: a scientific statement from the American Heart Association. Circulation. 2012 May 22;125(20):2520-44. doi: 10.1161/CIR.0b013e31825719f3. Epub 2012 Apr 18. PMID 22514251
- [Derived] Montenegro MM, Ribeiro IWJ, Kampits C, Saffi MAL, Furtado MV, Polanczyk CA, Haas AN, Rosing CK. Randomized controlled trial of the effect of periodontal treatment on cardiovascular risk biomarkers in patients with stable coronary artery disease: Preliminary findings of 3 months. J Clin Periodontol. 2019 Mar;46(3):321-331. doi: 10.1111/jcpe.13085. Epub 2019 Mar 6. PMID 30761568
- [Derived] Saffi MA, Furtado MV, Montenegro MM, Ribeiro IW, Kampits C, Rabelo-Silva ER, Polanczyk CA, Rosing CK, Haas AN. The effect of periodontal therapy on C-reactive protein, endothelial function, lipids and proinflammatory biomarkers in patients with stable coronary artery disease: study protocol for a randomized controlled trial. Trials. 2013 Sep 6;14:283. doi: 10.1186/1745-6215-14-283. PMID 24010954
- See also: School of Dentistry homepage — http://www.ufrgs.br/odonto
- See also: University Hospital homepage — http://www.hcpa.ufrgs.br